CLINICAL TRIAL: NCT06718465
Title: Development of Combined Imaging and Informatics Based Approaches to Understanding Cardiovascular Disease.
Brief Title: Integrated Informatics-imaging Approaches to Cardiovascular Disease.
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 152959
Record Dates: First submitted 2014-11-10; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-05

CONDITIONS: Atherosclerosis; Myocardial Infarction; Sudden Cardiac Death
MeSH Terms: conditions — Atherosclerosis; Myocardial Infarction; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At the time of autopsy sections of heart arteries, aortic valve and a sample of blood will be taken for gene and protein expression studies and further imaging studies.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sudden Cardiac Death Victim with coronary artherosclerosis: Sudden Death victims (>18 years old) who have died in the community and there is supportive evidence of myocardial infarction on autopsy.
- Sudden Death Victim without coronary artherosclerosis: Sudden Death victims (>18 years old) who have died in the community with no evidence of coronary atherosclerosis or myocardial infarction on autopsy.

SUMMARY:
Hardening of the arteries (atherosclerosis) is a common disorder that causes heart attacks. In the United Kingdom heart attacks are the commonest cause of death. Combined positron emission tomography (PET) and computer tomography (CT) scans are a new way of assessing atherosclerosis. Using the radiotracer 18F-Fluoride, this study proposes to perform combined PET CT scans on post-mortem hearts from participants with or without a history of heart disease. It will then be able to compare the hot spots found on these scans with what investigators can see under the microscope when looking at heart artery specimens, assess which genes are switched on and proteins present in the hot spots. This will give us an insight into what hot spots on PET CT scans are identifying in areas of atherosclerosis. It will also provide new information relating to the underlying processes that give rise to atherosclerosis and the development of heart attacks. This will pave the way for the future development of new treatments.

DETAILED DESCRIPTION:
Hardening of the arteries (atherosclerosis) is a very common health problem that can lead to fatal or disabling heart attacks or strokes. On many levels, it remains an incompletely understood illness.

Until relatively recently, the only way of assessing the severity of, or risk posed by, atherosclerosis was to measure the degree to which it narrowed a particular blood vessel. This method only tells part of the story; investigators now know that frequently the 'culprit area' of atherosclerosis that causes a heart attack or stroke doesn't necessarily result in narrowing of the blood vessel i.e. if investigators only measure narrowness they will miss lots of 'bad' atherosclerosis.

Combined PET CT scans not only provide more information about the composition and architecture of the atherosclerosis but can provide data about the processes (at the chemical and cellular level) that underlie the disease. Hardened arteries with areas of early calcification (deposits of calcium) are usually the culprits that lead to heart attacks. Early calcification can be detected using 18F-Fluoride PET CT scans. It has previously been described by the Chief Investigator and colleagues that hot spots on 18F-Fluoride PET CT scans are associated with rupture of hardened arteries in stroke patients.

The aim of this study is to explore whether hot spots on 18F-Fluoride PET CT scans are identifying early calcification in heart arteries and to use 18F-Fluoride PET CT imaging to gain a deeper insight into the progression of atherosclerosis. It is not feasible to perform detailed examinations of heart arteries in living patients. For this reason post-mortem examination of heart arteries offers a valuable opportunity to correlate PET CT scan findings with biological processes in order to get an understanding of what 'hot spots' on PET/CT scans are actually representing at the tissue level.

This study proposes to explore the biological processes in heart arteries identified with 18F-Fluoride PET CT imaging. Post-mortem hearts of patients both with and without a history of heart disease will be scanned to be able to define what is going on at the gene expression and protein level in the areas of 'hot spots' on CT PET scans.

ELIGIBILITY:
Inclusion Criteria:

* Sudden death victims dying in the community. Patients with or without a history of ischaemic heart disease.

Exclusion Criteria:

* Age under 18 years old. Suspicion around the cause of death, or cases of homicide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include sudden death victims who have died in the community.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
18F-fluoride uptake denotes microcalcification and atherosclerosis in aortic valves and coronary arteries | 2 years
  18F-fluoride uptake denotes microcalcification and atherosclerosis in aortic valves and coronary arteries and the pathways for gene and protein expression that are associated with this remain to be defined and this was assessed by PET/CT imaging